CLINICAL TRIAL: NCT04972994
Title: Surgical Outcomes After Laparoscopic Intracorporeal Versus Extracorporeal Anastomosis for Right and Left Hemicolectomies In Management of Colonic Cancers
Brief Title: Laparoscopic Colectomies In Management of Colonic Cancers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdullah Atyah Ali, Assistant lecture general surgery, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med206018
Record Dates: First submitted 2021-07-06; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Laparoscopic Colectomy; Cancer Colon; Intracorporeal Anastomosis
Keywords: laparoscopic; intracorporeal; extracorporeal; anastomosis; hemicolectomies; , colonic cance
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: right and left hemicolectomies in colonic cancers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic intracorporeal anastomosis for right and left hemicolectomies (Active Comparator): Surgical outcomes after laparoscopic intracorporeal versus for right and left hemicolectomies in management of colonic cancers
  Interventions: Procedure: laparoscopic intracorporeal versus extracorporeal anastomosis for right and left hemicolectomies
- laparoscopic extracorporeal anastomosis for right and left hemicolectomies (Active Comparator): Surgical outcomes after laparoscopic extracorporeal anastomosis for right and left hemicolectomies in management of colonic cancers
  Interventions: Procedure: laparoscopic intracorporeal versus extracorporeal anastomosis for right and left hemicolectomies

INTERVENTIONS:
Procedure: laparoscopic intracorporeal versus extracorporeal anastomosis for right and left hemicolectomies — laparoscopic intracorporeal versus extracorporeal anastomosis for right and left hemicolectomies in management of colonic cancers

SUMMARY:
The aim of this study is to compare the Surgical outcomes after laparoscopic intracorporeal versus extracorporeal anastomosis for right and left hemicolectomies in management of colonic cancers .

DETAILED DESCRIPTION:
This is clinical trial ,Interventional quasi experiment study to evaluate the surgical outcomes between intracorporeal versus extracorporeal anastomosis in laparoscopic right and left hemicolectomies including post operative pain, hospital stay, leakage from anastomosis, early recurrence, hernias patient satisfaction operative time and more surgical outcomes.

In Egyptian hospitals. Source of data the investigators follow up and medical reports and more . surgical procedures This trial including two groups of patients with right and left cancer colon undergoing Laparoscopic colectomy. First group (A) will be operated as intracorporeal anastomosis while the second group (B) will be operated as extracorporeal anastomosis.

Sample size more than 50 person Statistical analysis plan Statistical Package for the Social Sciences (SPSS) program

ELIGIBILITY:
Inclusion Criteria:

* Patients had to present histologically confirmed cancer( right and left) colon.
* All grades of cancer will be included.
* Cancer at cecum ,appendix, ascending colon, hepatic flexure or at splenic flexure , descending colon and sigmoid colon.

Exclusion Criteria:

* Locally advanced disease with invasion of adjacent important organs.
* Acute bowel obstruction or perforation from cancer.
* Pregnant ladies.
* Rectal cancer and transverse colon cancer.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
intraoperative time of surgery | intraoperative time of surgery
  intraoperative time of surgery by minutes
post operative hospital stay | up to 1 year
  post operative hospital stay by days
Post operative leakage | 1 year
  Post operative leakage of anastomosis by follow up ultrasound, Abdominal Xray erect & wound infection
early recurrence of the cancer | 6 months after surgery
  early recurrence of the cancer by CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Omar AS Al tabary, Professor, Study Director — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt